CLINICAL TRIAL: NCT02356198
Title: Exparel Transversus Abdominis Plane Block vs Intrathecal Analgesia In Colorectal Surgery: A Prospective Randomized Trial
Brief Title: Exparel Transversus Abdominis Plane Block vs Intrathecal Analgesia In Colorectal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Dorin T. Colibaseanu, M.D., PI, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14-003143
Record Dates: First submitted 2015-01-31; First posted 2015-02-05 (Estimated); Results first posted 2019-02-05 (Actual); Last update posted 2019-03-07 (Actual); Status verified 2019-03

CONDITIONS: Conditions Requiring Colorectal Surgery
MeSH Terms: interventions — Hydromorphone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TAP block (EXPAREL) (Active Comparator): After induction of anesthesia, the patients will receive a single injection with 133 mg of EXPAREL in the transversus abdominis plane (TAP), on each side, suspended in 20 milliliters (mL) of injectable saline.
  Interventions: Drug: EXPAREL
- Intrathecal opioid (IT) (Active Comparator): single injection intrathecal hydromorphone analgesia given preoperatively
  Interventions: Drug: Intrathecal hydromorphone

INTERVENTIONS:
Drug: EXPAREL — transversus abdominis plane injection
  Other Names: liposomal bupivacaine
  Arms: TAP block (EXPAREL)
Drug: Intrathecal hydromorphone — Intrathecal opioid administration
  Other Names: dilaudid
  Arms: Intrathecal opioid (IT)

SUMMARY:
This study is prospective, randomized trial in which EXPAREL TAP block is compared to standard IT opioid administration, in relieving postoperative pain, decreasing length of stay, and use of narcotic medication.

DETAILED DESCRIPTION:
Primary Objective To assess efficacy of EXPAREL TAP blocks in improving pain scores for 48 hours postoperatively, and in reducing total oral morphine equivalents (OME) use, compared to standard Intrathecal opioid administration (IT).

Secondary Objective Assess the length of stay (LOS), postoperative ileus (POI) incidence, and the use of intravenous patient controlled analgesia (PCA) in patients that had EXPAREL TAP blocs compared to IT.

ELIGIBILITY:
Inclusion Criteria:

* • All patients undergoing elective laparoscopic or open colorectal resections who are eligible for IT

  * Age >18 years
  * BMI <40
  * Ability to understand and read English

Exclusion Criteria:

* • Not able or unwilling to sign consent.

  * Currently pregnant or lactating.
  * Patients with chronic pain, requiring daily opiate use at time of surgery.
  * Patients intolerant of opiates, NSAIDS, acetaminophen or local anesthetics.
  * Patients requiring emergent surgery.
  * Abdominoperineal resections
  * Any contraindications to neuraxial analgesia (coagulopathy, localized infection at the potential site of injection, pre-existing spinal canal pathology)
  * Patients with a diagnosis of inflammatory bowel disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 209 (Actual)
Dates: Start 2015-03; Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dorin Colibaseanu, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Florida, Jacksonville, Florida, United States

REFERENCES:
- [Derived] Colibaseanu DT, Osagiede O, Merchea A, Ball CT, Bojaxhi E, Panchamia JK, Jacob AK, Kelley SR, Naessens JM, Larson DW. Randomized clinical trial of liposomal bupivacaine transverse abdominis plane block versus intrathecal analgesia in colorectal surgery. Br J Surg. 2019 May;106(6):692-699. doi: 10.1002/bjs.11141. Epub 2019 Mar 28. PMID 30919948
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | TAP Block (EXPAREL) | Intrathecal Opioid (IT)
Started | 104 | 105
Completed | 102 | 98
Not Completed | 2 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TAP Block (EXPAREL) | Intrathecal Opioid (IT) | Total
Number analyzed (Participants) | 102 | 98 | 200
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 61 [50 to 68] | 58 [49 to 69] | 60 [49 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 43 | 88
  Male | 57 | 55 | 112
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 102 | 98 | 200

OUTCOME MEASURES:

1. Primary Outcome: Mean Pain Score
Description: Postoperative mean pain score for 48 hours after surgery. Pain was assessed on a 0 to 10 point visual analog scale (VAS), with 0 indicating no pain and 10 indicating severe pain. The mean pain score was summarized as the area under the curve (AUC) of the observed pain score, normalized for the total time of observation.
Time Frame: First 48 hours post operative
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | TAP Block (EXPAREL) | Intrathecal Opioid (IT)
Number analyzed (Participants) | 102 | 98
score on a scale | 3.0 [2.7 to 3.3] | 2.4 [2.1 to 2.7]
Statistical Analysis 1: Comparison: TAP Block (EXPAREL) vs Intrathecal Opioid (IT); Test type: Superiority; p = 0.007, t-test, 2 sided

2. Primary Outcome: Total Morphine Milligram Equivalents Use (MME)
Description: The total cumulative use of opioids administered within 48 hours after surgery. MME is a standard value based on morphine and its potency assigned to all opioids to represent relative potencies.
Time Frame: First 48 hours post operative
Measure: Median (95% Confidence Interval); unit: total morphine milligram equivalents
Arm/Group | TAP Block (EXPAREL) | Intrathecal Opioid (IT)
Number analyzed (Participants) | 102 | 98
total morphine milligram equivalents | 47.5 [35.6 to 65.9] | 32.5 [24.4 to 42]
Statistical Analysis 1: Comparison: TAP Block (EXPAREL) vs Intrathecal Opioid (IT); Test type: Superiority; p = 0.102, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Total Length of Hospital Stay
Description: Length of stay was defined as the total number of nights spent in the hospital after surgery.
Time Frame: post-operative to discharge
Measure: Median (95% Confidence Interval); unit: nights
Arm/Group | TAP Block (EXPAREL) | Intrathecal Opioid (IT)
Number analyzed (Participants) | 102 | 98
nights | 3 [3 to 3] | 3 [3 to 4]
Statistical Analysis 1: Comparison: TAP Block (EXPAREL) vs Intrathecal Opioid (IT); Test type: Superiority; p = 0.85, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Number of Participants With Post-operative Ileus
Description: Post-operative ileus was defined as the inability to tolerate oral diet and/or the absence of flatus over 24 hours after surgery.
Time Frame: 24 hours post-operatively
Measure: Count of Participants; unit: Participants
Arm/Group | TAP Block (EXPAREL) | Intrathecal Opioid (IT)
Number analyzed (Participants) | 102 | 98
Participants | 11 | 14
Statistical Analysis 1: Comparison: TAP Block (EXPAREL) vs Intrathecal Opioid (IT); Test type: Superiority; p = 0.454, Chi-squared

5. Secondary Outcome: Use of Intravenous Patient-controlled Analgesia
Description: The total number of patients that used patient-controlled analgesia within 48 hours after surgery.
Time Frame: First 48 hours post-operative
Measure: Count of Participants; unit: Participants
Arm/Group | TAP Block (EXPAREL) | Intrathecal Opioid (IT)
Number analyzed (Participants) | 102 | 98
Participants | 5 | 1
Statistical Analysis 1: Comparison: TAP Block (EXPAREL) vs Intrathecal Opioid (IT); Test type: Superiority; p = 0.212, Fisher Exact

ADVERSE EVENTS:
Time Frame: The study treatment follow-up period was defined as 30 days +/- 10 days following the last administration of study treatment.
Arm/Group | TAP Block (EXPAREL) | Intrathecal Opioid (IT)
All-Cause Mortality (participants affected / at risk) | 0/102 | 0/98
Serious Adverse Events (participants affected / at risk) | 4/102 | 4/98
Other Adverse Events (participants affected / at risk) | 0/102 | 0/98
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TAP Block (EXPAREL) (N=102) | Intrathecal Opioid (IT) (N=98)
Peristomal wound infection (Infections and infestations) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Spinal fluid leakage (Nervous system disorders) | 0 (0) | 1 (1)
Bleeding at injection site (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Intra-abdominal abscess (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anastomosis leakage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Tachypnea with hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-02): https://cdn.clinicaltrials.gov/large-docs/98/NCT02356198/Prot_SAP_000.pdf